CLINICAL TRIAL: NCT06056661
Title: Culturally Adapting Individually-oriented Relationship Education (Within My Reach) for Latino Sexual Minority Men
Brief Title: Within My Reach (WMR) Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Mental Research Institute (Other)
Responsible Party: Principal Investigator, Audrey Harkness, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20221114
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hiv; Violence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WMR group (Experimental): Participants in this group will receive the WMR program for up to 5 weeks.
  Interventions: Behavioral: WMR

INTERVENTIONS:
Behavioral: WMR — Participants will complete up to five sessions that will take 2 hours each. Sessions will take place in person. Participants will learn skills related to getting into and out of romantic relationships and identifying and pursuing goals for romantic relationships.

SUMMARY:
The purpose of this study is to adapt a relationship education program. The research team is adapting so that it is helpful for Latino sexual minority men.

ELIGIBILITY:
Inclusion:

* Identify as Latino/e/x or Hispanic
* Age 18 years or older
* Currently reside in Miami-Dade County or Broward County
* Identify as gay, bisexual, or other non-heterosexual identity
* Identify as a man
* Comfortable speaking English

Exclusion:

* Unable to provide consent
* Deemed that participating would be potentially harmful to the participant or research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as a man
Enrollment: 16 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Acceptability, as measured by the Acceptability of Intervention Measure (AIM) | Up to 3 months
  The AIM consists of four questions that assess acceptability. Responses range from 1 (completely disagree) to 5 (completely agree). Scales are created by averaging responses.
Appropriateness, as measured by the Intervention Appropriateness Measure (IAM) | Up to 3 months
  The IAM consists of four questions that assess appropriateness. Responses range from 1 (completely disagree) to 5 (completely agree). Scales are created by averaging responses.

SECONDARY OUTCOMES:
Change in Sexual Risk Composite, as measured by HIV risk assessment | Baseline compared to up to 3 months
  Participants will answer questions about engagement in anal or vaginal sex, sexual partners' HIV status, current pre-exposure prophylaxis (PrEP) use and adherence (if HIV-negative or unknown HIV status), viral load (if living with HIV), A composite score will be calculated to determine whether or not the participant engaged in sexual behavior that could lead to HIV transmission or acquisition. A score of 1 means that the participant engaged in sexual behavior that could lead to HIV acquisition or transmission. A score of 0 means that they did not.
Change in Acceptance of Couple Violence | Baseline compared to up to 3 months
  The outcome will be measured with the five-item general violence subscale from the Acceptance of Couple Violence Scale. The items will be rated on a scale from 1 (strongly disagree) to 4 (strongly agree). Scales are created by averaging responses.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Harkness, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No